CLINICAL TRIAL: NCT00302887
Title: Short and Long Term Results of Connective Tissue Manipulation and Combined Ultrasound Therapy in Patients with Fibromyalgia
Brief Title: Connective Tissue Manipulation and Combined Ultrasound Therapy in Patients with Fibromyalgia
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, İlkim Çıtak Karakaya, Research Assistant, Hacettepe University
Other Study IDs: HEK06/12-39
Record Dates: First submitted 2006-03-14; First posted 2006-03-15 (Estimated); Last update posted 2025-03-14 (Actual); Status verified 2006-03

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; connective tissue manipulation; ultrasound therapy; high voltage pulsed galvanic stimulation
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Device: combined ultrasound therapy
Procedure: connective tissue manipulation

SUMMARY:
The aim of this study was to evaluate the short term and one year follow-up results of connective tissue manipulation and combined ultrasound therapy (ultrasound and high voltage pulsed galvanic stimulation) in terms of pain, complaint of non-restorative sleep and impact on the functional activities in patients with fibromyalgia.

DETAILED DESCRIPTION:
This is an observational prospective cohort study, investigating short and long term results of physiotherapy applications in 20 female patients with fibromyalgia. Physical characteristics of the subjects were recorded. Intensity of pain, complaint of non-restorative sleep, and impact of fibromyalgia on functional activities were evaluated by visual analogue scales. All evaluations were performed before and after 20 sessions of treatment, which included connective tissue manipulation of the back daily, for a total of 20 sessions and combined ultrasound therapy of the upper back region every other session. One year follow-up evaluations could be performed on 14 subjects.

ELIGIBILITY:
Inclusion Criteria:

Women with pain depending to FM, with an intensity interfering to activities of daily living for a duration of at least six months, able to participate of 20 physiotherapy sessions within a four week period, volunteer for participating to the study without taking any drugs acting on the nervous system such as antidepressants, myorelaxants, analgesics or hypnotics, in the study period.

Exclusion Criteria:

evidence of neurological, infectious, endocrine and other inflammatory rheumatic diseases, and experience with any kind of manual and/or electrotherapy, within six months before the study.

Ages: 19 Years to 68 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample was derived from a population of 83 FM outpatients of the Hacettepe University School of Physical Therapy and Rehabilitation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2003-08 (Actual); Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
pain intensity | All evaluations were performed before and after 20 sessions of treatment.
  The intensity of pain was evaluated by 0-10 cm visual analogue scales (VASs). On the VAS, "0" indicated "no pain" and the "10" indicated "the worst imaginable pain".

CONTACTS AND LOCATIONS:
Overall Officials: İlkim Çıtak Karakaya, PT. PhD., Principal Investigator — PT. PhD. Assist. Prof.; Türkan Akbayrak, PT. PhD., Study Director — PT. PhD. Assoc. Prof.; Funda Demirtürk, PT. PhD., Study Chair — Research assistant; Gamze Ekici, PT. MSc., Study Chair — Research assistant; Yeşim Bakar, PT. PhD., Study Chair — Assist. Prof.
Locations (1):
- Hacettepe University, School of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)